CLINICAL TRIAL: NCT06706193
Title: Wear Resistance of Highly Crosslinked Cemented Polyethylene Cups in Young Patients
Brief Title: HXLPE Vs CPE Cups Under 50 Years
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HXLPE_50y
Record Dates: First submitted 2024-11-21; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Osteoarthritis, Hip
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Intervention Model Description: After obtaining informed consent, the participants were randomized to a surgical intervention with the use of 60 sealed envelopes which were opened by the surgeon in theatre just before surgery.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Active Comparator)
  Interventions: Procedure: Total hip arthroplasty using CPE
- Intervention group (Experimental)
  Interventions: Procedure: Total hip arthroplasty using HXLPE

INTERVENTIONS:
Procedure: Total hip arthroplasty using CPE
  Arms: Control group
Procedure: Total hip arthroplasty using HXLPE
  Arms: Intervention group

SUMMARY:
This randomized controlled trial evaluated the long-term wear of cemented highly cross-linked polyethylene (HXLPE) versus conventional polyethylene (CPE) acetabular cups in patients under 50 years undergoing primary total hip arthroplasty (THA).

All surgeries were performed at Radboud University Medical Center by three surgeons using a posterolateral approach. Acetabular components included either highly cross-linked polyethylene (HXLPE) cups (X3 RimFit) or conventional polyethylene (CPE) cups (Exeter Contemporary Flanged). Both were implanted with bone cement, and femoral components consisted of Exeter V40 stems with 28 mm cobalt-chromium heads. Impaction bone grafting (IBG) was routinely used, with mesh applied in cases of acetabular bone defects.

Radiographs were taken preoperatively and at 10-year follow-up using standardized protocols. Polyethylene wear was assessed with PolyWare software, creating 3D models from baseline and 10-year radiographs to calculate linear and volumetric wear. Cup inclination and osteolysis were evaluated in three acetabular zones (DeLee and Charnley classification).

ELIGIBILITY:
Inclusion Criteria:

* primary THA
* age under 50 years

Exclusion Criteria:

* THA due to an oncological condition

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 59 (Actual)
Dates: Start 2010-10-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Linear wear (mm/y) | 10 years
Volumetric wear (mm3/y) | 10 years

SECONDARY OUTCOMES:
Cup survival (%) | 10 years

IPD SHARING:
Plan to Share IPD: Undecided